CLINICAL TRIAL: NCT02720770
Title: Proposition Pour un Traitement Par Hormone de Croissance Des Enfants Atteints de Rachitisme Hypophosphatemique Familial
Brief Title: Growth Hormone Treatment in Children With Hypophosphatemic Rickets
Acronym: GH-XLH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Alessia Usardi, Professor, Bicetre Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBM 03-47
Record Dates: First submitted 2016-03-15; First posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: X Linked Hypophosphatemic Rickets
Keywords: growth hormone
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- norditropine simplex (Experimental)
  Interventions: Drug: norditropine simplex

INTERVENTIONS:
Drug: norditropine simplex
  Other Names: growth hormone

SUMMARY:
This study evaluates the effect on height of a two year treatment with growth hormone in 19 children with X linked hypophosphatemic rickets.

ELIGIBILITY:
Inclusion Criteria:

* clinical, biochemical and genetic diagnosis of XLH
* height SDS < 2
* at least two years of treatment with oral phosphate and calcitriol

Exclusion Criteria:

* uncontrolled rickets (ALP>600 IU)
* growth hormone deficiency
* hyperparathyroidism, nephrocalcinosis, renal insufficiency
* associated disease
* previous treatment with growth hormone

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
change from baseline in height SDS (standard deviation score) | at year one and year two from baseline

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rothenbuhler A, Esterle L, Gueorguieva I, Salles JP, Mignot B, Colle M, Linglart A. Two-year recombinant human growth hormone (rhGH) treatment is more effective in pre-pubertal compared to pubertal short children with X-linked hypophosphatemic rickets (XLHR). Growth Horm IGF Res. 2017 Oct;36:11-15. doi: 10.1016/j.ghir.2017.08.001. Epub 2017 Aug 15. PMID 28822957